CLINICAL TRIAL: NCT05658848
Title: Effect of Collaborative Infertility Counseling on Coping Strategies and Marital Satisfaction Among Women Undergoing in Vitro Fertilization: A Randomized Control Trial
Brief Title: Effect of Collaborative Infertility Counseling on Coping Strategies and Marital Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Port Said University (Other)
Collaborators: Mansoura University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Abdelsattar Zoromba, Principal Investigator, Port Said University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P.0335
Record Dates: First submitted 2022-12-09; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Fertility Issues
MeSH Terms: conditions — Infertility | interventions — Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women cases (Experimental)
  Interventions: Other: Collaborative infertility counseling
- women control (No Intervention)

INTERVENTIONS:
Other: Collaborative infertility counseling — Collaborative infertility counseling for coping stratigies and marital satisfaction
  Other Names: Counseling
  Arms: women cases

SUMMARY:
Effect of collaborative infertility counseling on coping strategies and marital satisfaction among women undergoing in vitro fertilization: a randomized control trial

ELIGIBILITY:
This study will include a non-probability purposive sample of 136 infertile women undergoing IVF recruiting from the outpatient clinics according to the following inclusion criteria:

* age 20 to 45 years
* having a general health score below 28,
* can read and write,

Exclusion criteria include:

* psychiatric problems,
* previous assisted reproductive technology failure,
* leave the intervention for any reason and
* women suddenly experience severe traumatic or psychological events.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Coping strategies | Three Months
  The Ways of Coping-Revised (WOC-R) questionnaire will be adopted from Folkman, Lazarus, Pimley, & Novacek, (1987) to evaluate women coping styles. It contains 31 items and 8 subscales graded by a 3-point Likert scale. It is divided into problem-focused and emotion-focused coping strategies. The problem-focused strategy includes 4 subscales: planful problem solving, seeking social support, accepting responsibility, and positive reappraisal. The emotional-focused coping strategy includes 4 subscales: confrontive coping, self-controlling, distancing, and escape/avoidance. The responses will be rated on a 3-point scale (0 = didn't use to 2 = used all the time).
Marital Satisfaction | Three Months
  The Marital Satisfaction Index (MSI) was developed by Cheung & Hudson, (1982) to measure the degree of marital satisfaction. It consists of 25 items of which 13 are positively worded and 12 are negatively worded. The responses will be rated on a 5-point Likert scale (1 = None of the time, 2 = Very rarely, 3 = Sometimes, 4 = Most of the time, and 5 = All the time). The minimum and maximum scores of the MSI are 25 and 75, respectively. The higher score (above 30) indicates women's dissatisfaction. The GHQ-28 and FPI will be used to assess women's general health and perceived fertility-related stress respectively (Goldberg & Hillier, 1979; Sherrard, Newton, & Glavac, 1999).

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University hospitals, Al Mansurah, Egypt